CLINICAL TRIAL: NCT05534230
Title: Is Dexmedetomidine Effective at Reducing Pain Scores and Opioid Consumption in Coronary Artery Bypass Grafting (CABG) Patients
Brief Title: Dexmedetomidine for Pain Reduction in CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Sandeep Krishnan, Associate Professor of Anesthesiology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-012-SJMO
Record Dates: First submitted 2022-08-28; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Analgesia
Keywords: Dexmedotimidine, CABG, Pain Management
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This Study will be consist of two arms one treatment arm and one control arm.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Intravenous normal saline at a standard dose of 0.5mcg/kg/hr continued to postop until extubation.
  Interventions: Drug: Saline
- Dexmedotimidine Group (Active Comparator): Intravenous dexmedetomidine infusion started after induction at a standard dose of 0.5mcg/kg/hr and continued until extubation.
  Interventions: Drug: Dexmedetomidine Injectable Solution

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Solution — Intravenous dexmedetomidine infusion started after induction at a standard dose of 0.5mcg/kg/hr and continued until extubation.
  Other Names: Precedex, Hospira
  Arms: Dexmedotimidine Group
Drug: Saline — Intravenous normal saline at a standard dose of 0.5mcg/kg/hr continued to postop until extubation.
  Other Names: solution of Sodium Chloride
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether adjuvant intravenous dexmedetomidine infusion starting after induction of general anesthesia can provide superior pain management (decrease pain scores) and decrease opioid administration, without increasing nausea/vomiting, compared to patients receiving only opioid and acetaminophen for the patients which going through coronary artery bypass grafting (CABG)?

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) involves a median sternotomy and subsequent surrounding surgical dissection. Resulting tissue damage can lead to neurogenic inflammation and release of inflammatory mediators that promote acute postoperative pain . Given the location of the incision, uncontrolled acute postoperative pain after CABG can be associated with significant pulmonary complications . Additionally, acute pain activates the sympathetic nervous system which can have deleterious effects on multiple organ systems including the cardiovascular, gastrointestinal, and endocrine systems .

Dexmedetomidine is a sympatholytic agent acting on the alpha2 adrenergic receptor. It was originally used as an anxiolytic and sedative agent perioperatively and in the intensive care unit (ICU) by decreasing adrenergic response in the locus coeruleus and, thus, indirectly increasing gamma-aminobutyric acid (GABA) neurons downstream .

The use of perioperative dexmedetomidine has expanded; it has been studied as part of multimodal analgesic regimens as well as an adjuvant analgesic agent. It can directly work on the peripheral nervous system and inhibit C fibers and Aδ fibers to attenuate peripheral transmission of nociception . Within the central nervous system, dexmedetomidine inhibits adrenergic nociception transmission from the locus coeruleus through the spinal cord, which in turn prevent the release of nociceptive neurotransmitters and biochemicals at the presynaptic membrane . Also, alpha receptor agonism at the presynaptic membrane inhibits the release of norepinephrine and prevents nociceptive signals to the brain . Given its action at multiple sites within the nociceptive pathway, dexmedetomidine can be administered via various modalities including intravenous, intramuscular, neuraxial, peripheral nerve block, and topical.

Given its sympatholytic effect, reported side effects of dexmedetomidine are hypotension and bradycardia. In a meta-analysis of the safety of dexmedetomidine in cardiac surgery patients done by Wang et al., there was 3.4 times increased incidence of bradycardia with patients on dexmedetomidine compared to the control; however, there was no statistically significant difference in hypotension . Bradycardia occurs more often when dexmedetomidine is infused at 0.75-1 mcg/kg/hr than at 0.5mcg/kg/hr . The meta-analysis included publications that incorporated a loading dose prior to an infusion at a set dose; high plasma level of dexmedetomidine has been associated with cross reactivity with alpha1 stimulation and subsequent vasoconstriction resulting in hypertension and reflex bradycardia. However, elimination of the loading dose has been shown to eliminate the hemodynamic effect . Any intraoperative bradycardia or hypotension can be treated with anticholinergics and vasoactive agents, respectively, without postoperative bradycardia, hypotension, or related complications .

Compared to conventional opioid analgesia for acute postoperative pain, dexmedetomidine analgesia has limited adverse impact on the cardiovascular, pulmonary, and gastrointestinal systems . Perioperative dexmedetomidine has consistently demonstrated improved acute postoperative pain and reduced narcotic requirement in noncardiac surgeries including open and laparoscopic abdominal, open and laparoscopic gynecological, and neuro surgeries compared to traditional opioid therapy .

Previous research has shown great benefits of perioperative dexmedetomidine use in cardiac surgery patients. During open heart surgery, exposure of blood to the cardiopulmonary bypass (CPB) circuit and ischemia-reperfusion of organs contribute to a surge of cytokines and other inflammatory mediator. Dexmedetomidine reduces the circulating plasma level of proinflammatory cytokines, norepinephrine, and cortisol after cardiac surgery with CPB .

Acute kidney injury (AKI) is one of the more common complications of open-heart surgery and CPB. Multiple etiologies play a role in the pathophysiology, including reduced perfusion during aortic cross clamping, possible blood product transfusion, and generalized inflammatory state during CPB. In a meta-analysis done by Peng et al. involving nine studies, the incidence of AKI was reduced in patients receiving dexmedetomidine infusion, most significantly when started preoperative or intraoperative with or without postoperative continuation .

In another meta-analysis done by Li et al. that included fifteen studies and 2813 patients, postoperative delirium was reduced in patients receiving perioperative dexmedetomidine. Interestingly, they also did not find any statistically significant difference in hypotension or bradycardia. Perioperative dexmedetomidine also demonstrated reduction in in-hospital mortality, 30 day mortality, and 1 year mortality and overall incidence of any postoperative complications in cardiac surgery . Dexmedetomidine in animal models has shown to protect the myocardium from ischemia by increasing adenosine-induced coronary vasodilation and provide myocardial preconditioning to attenuate myocardial ischemia-reperfusion injury ; however, clinical data on human subjects are inconclusive.

Currently, there is limited data and literature on the role of perioperative dexmedetomidine on acute post-operative pain in cardiac surgery patients. No studies have been done on the relationship between dexmedetomidine infusion that has been started after induction of general anesthesia continued until extubation and acute post-operative pain in CABG with CPB patients.

At SJMO, patients who undergo CABG currently receive intraoperative intravenous fentanyl and postoperative oral acetaminophen and intravenous and oral opioids for perioperative pain control.

The purpose of this study is to determine whether adjuvant intravenous dexmedetomidine infusion starting after induction of general anesthesia can provide superior pain management (decrease pain scores) and decrease opioid administration, without increasing nausea/vomiting, compared to patients receiving only opioid and acetaminophen.

Hypothesis: There is a significant difference in the VAS pain scores, number of VAS score greater than 5, rate of opioid consumption (postop and intraop), and the percentage of with PONV, for patients having CABG with continuous intravenous infusion of dexmedetomidine after induction of general anesthesia.

Null: There is no significant difference in the VAS pain scores, number of VAS score greater than 5, rate of opioid consumption (postop and intraop), and the percentage of patience with PONV, for patients having CABG with continuous infusion of dexmedetomidine after induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be between 18 years old and 100 years old. Both men and women will be eligible for this study. We will aim to have approximately 50% men and 50% women. People of all races and ethnic origins are eligible.

Patients should be undergoing CABG (coronary artery bypass grafting ) under general anesthesia with CPB (Cardiopulmonary bypass).

Exclusion Criteria:

Patients will be excluded who are receiving valve replacement with CABG, Class I emergent CABG, receiving regional anesthesia, clinically significant preoperative neurologic, cardiac, pulmonary, renal, or hepatic disease that cannot tolerate dexmedetomidine infusion, or reported allergy to dexmedetomidine. People taking chronic opioid will also be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-06 (Estimated); Primary Completion 2023-07-10 (Estimated); Study Completion 2024-05-09 (Estimated)

PRIMARY OUTCOMES:
Visual analog pain (VAS) scores at 6, 12, 18, and 24 hours post-surgery | measured at 6, 12, 18, and 24 hours post-surgery
  Pain scores are measured by asking the patients to rank their pain from 1 to 10
Total opioid consumption in the first 24 hours after surgery (Oral morphine equivalents) | 24 Hours post surgery
  the totalOral morphine equivalent dose of Opioids received by the patient 24 hour after the surgery is calculated

SECONDARY OUTCOMES:
Incidence of post-operation nausea and vomiting (PONV) (treatment with anti-emetic) in the first 24 hours | 24 Hours Post Surgery
  Incidence of Nausea and/or Vomiting. This is a categorical variable with Yes and No answer for each patient
Incidence of pruritus (Percent of patients) | 24 hours Post Surgery
  This is a categorical variable with Yes and No answer for each patient
Total Acetaminophen intake | 24 Hours post surgery
  All the acetaminophen which is given to the patient is added as total mg
Total NSAID intake | 24 hours Post Surgery
  All the NSAID which is given to the patient is added as total mg
Incidence of atrial fibrillation | during Hospital Stay
  the incidence of atrial fibrillation which is is an irregular and often very rapid heart rhythm (arrhythmia) is recorded as YES or NO
Postoperative AKI based on AKIN | during Hospital Stay
  Criteria based on lab values from the morning of POD2 (>0.3 serum creatinine OR >150-200% from baseline OR UOP< 0.5mL/kg/hr for >6hours). Most patients meet RIFLE criteria within the first 48hours.
Vasoplegia | during Hospital Stay
  after coming off of cardiopulmonary bypass (hypotension with SVR<800 and CI > 2.2L/kg)- requiring more than 1 pressors
Hospital length of Stay | During Hospital Stay
  The duration of stay in ICU is recorded.
Incidence of intraop bradycardia | During Surgery
  (HR<40BPM or bradycardia requiring treatment)
Incidence of intraop hypotension | During Surgery
  (MAP <45/50mmHg AND requiring treatment)- during the entire case measuring how many "yes"
Hospital Length of Stay | During Hospital Stay
  The Duration of stay in Hospital is recorded

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zubrzycki M, Liebold A, Skrabal C, Reinelt H, Ziegler M, Perdas E, Zubrzycka M. Assessment and pathophysiology of pain in cardiac surgery. J Pain Res. 2018 Aug 24;11:1599-1611. doi: 10.2147/JPR.S162067. eCollection 2018. PMID 30197534
- [Background] Tang C, Xia Z. Dexmedetomidine in perioperative acute pain management: a non-opioid adjuvant analgesic. J Pain Res. 2017 Aug 11;10:1899-1904. doi: 10.2147/JPR.S139387. eCollection 2017. PMID 28860845